CLINICAL TRIAL: NCT01376960
Title: Ankle Block Versus Popliteal Fossa Block as Primary Anesthesia for Forefoot Surgical Procedures: A Prospective Comparison
Brief Title: Ankle Block Versus Popliteal Fossa Block as Primary Anesthesia for Forefoot Surgical Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121809A
Record Dates: First submitted 2009-07-29; First posted 2011-06-20 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Anesthesia; Forefoot Surgery
Keywords: forefoot surgery; Ankle Block; Popliteal Fossa Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single shot popliteal fossa block (Active Comparator)
  Interventions: Procedure: elective forefoot surgery
- ankle blocks (Active Comparator)
  Interventions: Procedure: elective forefoot surgery

INTERVENTIONS:
Procedure: elective forefoot surgery — Includes both soft-tissue and osseous procedures.

SUMMARY:
The purpose of this study is to compare, for the first time ever, single shot popliteal fossa blocks to ankle blocks as primary anesthesia for patients undergoing forefoot procedures. The primary outcome variable for this study is the percentage of patients that convert to general anesthesia following either a single shot popliteal fossa block or ankle block.

H0: There is no difference in the percentage of patients that convert to general anesthesia between single shot popliteal fossa blocks and ankle blocks.

HA: There will be a lower percentage of patients receiving a single shot popliteal fossa block that convert to general anesthesia compared to patients receiving an ankle block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective forefoot surgery, including both soft-tissue and osseous procedures

Exclusion Criteria:

* Diabetes
* Any form of Peripheral neuropathy
* Known allergy to local anesthesia
* Active infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Conversion to general anesthesia following either a single shot popliteal fossa block or ankle block | Participants will be followed for the duration of the surgery, an expected average of 2 hours
  Popliteal fossa and ankle blocks are types of anesthesia used during surgery. If these methods are not effective as an anesthetic during surgery the anethesiologist will convert to general anesthesia.

SECONDARY OUTCOMES:
Visual Analog Pain Scale (VAS) | 24 hours postoperatively
Patient Satisfaction | 48 hours postoperative
Length of Post Anesthesia Care Unit (PACU) stay | Up to 6 hours postoperative
  Length of PACU stay is calculated from the time the patient is taken from the operative suite to PACU, ie recovery, to the time the patient leaves PACU.
Narcotic Use | Up to 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Cohen, MD, Principal Investigator — OrthoCarolina, PA
Locations (1):
- OrthoCarolina, PA, Charlotte, North Carolina, United States